CLINICAL TRIAL: NCT02804997
Title: Evaluation of the Alveolar Recruitment Obtained During Non-invasive Ventilation After Cardiac Surgery
Acronym: ARCTICS
Status: Terminated | Type: Observational
Why Stopped: internal recruitment difficulties and reorganization of the Intensive Care Units
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2014_843_0020
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Thoracic Surgery
Keywords: non-invasive ventilation; cardiac surgery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
The great majority of cardiac surgery patients develop a degree of post-operatory respiratory failure. This is due to several factors. The predominant element in the onset of this respiratory impairment is the constitution of foci of pulmonary atelectasis, caused by peroperative hypoventilation (in the presence or absence of ECC). The incidence has been evaluated at between 54% and 92%, depending on the study. The use of NIV (non-invasive ventilation) might (through the application of continuous positive expiratory pressure) help to counter the development of these atelectasic foci.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* in the post-operative phase after elective cardiac surgery for aortic or mitral valve replacement, coronary revascularization or mixed surgery, hypoxemia or hypercapnia, with an indication for NIV,
* hemodynamic stability
* prior consent
* spontaneous ventilation
* social security coverage.

Exclusion Criteria:

* Under-18 patients
* complex cardiac surgery
* pregnancy
* pre-existing chronic obstructive respiratory disease (COPD > stage II)
* legal guardianship
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in the post-operative phase after elective cardiac surgery for aortic or mitral valve replacement, coronary revascularization or mixed surgery, hypoxemia or hypercapnia, with an indication for NIV, hemodynamic stability, prior consent, spontaneous ventilation, social security coverage
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

PRIMARY OUTCOMES:
Quantitative evaluation by thoracic CT scan | 3 hours
  Quantitative evaluation performed by thoracic CT scan of alveolar recruitment induced by NIV after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elie ZOGHEIB, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France